CLINICAL TRIAL: NCT06630052
Title: Incidence of Tenderness Opposite to Adductor Canal in Patients Suffering From Osteoarthritis Knee Pain. A Cohort Study.
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Abeer Ahmed, MD, Professor, Cairo University
Other Study IDs: MS-310-2023
Record Dates: First submitted 2024-01-31; First posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Knee Arthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: adductor canal clinical examination — clinical examination of the adductor canal in patients with knee pain not matching the radiological changes

SUMMARY:
Knee osteoarthritis (KOA) is a common knee disorder. The pathological changes affecting the knee are typically examined by using X-ray imaging to assess the narrowing of the joint space and the presence of osteophytes. However, some previous clinical trials have revealed a discrepancy between the severity of joint pain and the image finding even with the use of knee MRI. Some studies have revealed that there are age-related changes in the type of fibers with the formation of a network of transverse fiber bands, and this may cause some compression or traction on the neurovascular content of the adductor canal. Other studies noted the presence of excessive yellow-colored adipose tissue that stretches or entangles some nerve fibers. The primary outcome of this study will be the incidence rate of tenderness over the midthigh corresponding to the AC in patients with KOA who are complaining of severe pain that is discordant with the radiological finding.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with confirmed KOA by symptomatic (rated knee pain > four on a 10-point numeric rating pain scale (NRP scale)) and radiologically (Kellgren-Lawrence grades I, II ) findings

Exclusion Criteria:

* Post-traumatic knee osteoarthritis, oncological diseases, endocrine diseases (gout, diabetes), autoimmune diseases (rheumatoid arthritis), infectious diseases and patients with a history of previous knee surgeries or endoscopies

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients with confirmed KOA by symptomatic (rated knee pain > four on a 10-point numeric rating pain scale (NRP scale)) and radiologically (Kellgren-Lawrence grades I, II ) findings
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-08-15 (Actual); Study Completion 2024-09-15 (Actual)

PRIMARY OUTCOMES:
incidence of tenderness corresponding to the AC in patients complaining of severe pain with discordant with the radiological finding | time of clinical examination at the date of the visit to the pain clinic till the knee interventions up to 2 days
  the presence of tenderness by hand pressing over AC for 3-4 cm depth

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Abeer Ahmed Mohamed, Maadi, Cairo Governorate
  - Anesthesia department - Faculty of medicine- Cairo University, Cairo

IPD SHARING:
Plan to Share IPD: Undecided